CLINICAL TRIAL: NCT00183573
Title: HIV Prevention for STD Clinic Patients
Brief Title: HIV Prevention Program for Patients Receiving Care at a Sexually Transmitted Diseases Clinic
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of Rochester (Other); Syracuse University (Other)
Responsible Party: Principal Investigator, Michael P. Carey, Director, CBPM, The Miriam Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01MH068171 (NIH); R01MH068171 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2013-06-07 (Estimated); Status verified 2013-06

CONDITIONS: HIV Infections; Sexually Transmitted Diseases
Keywords: STDs; Sexual Behavior; Health Behavior; HIV Seronegativity
MeSH Terms: conditions — HIV Infections; Sexually Transmitted Diseases; Sexual Behavior; Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1 (Experimental): Brief Motivational Intervention only
  Interventions: Behavioral: Brief Motivational Intervention
- 2 (Experimental): Brief Informational Intervention only
  Interventions: Behavioral: Brief Informational Intervention
- 3 (Experimental): Brief Motivational Intervention + Intensive Informational Intervention
  Interventions: Behavioral: Brief Motivational Intervention; Behavioral: Intensive Informational Intervention
- 4 (Experimental): Brief Motivational Intervention + Intensive Information-Motivation-Behavioral Skills Intervention
  Interventions: Behavioral: Brief Motivational Intervention; Behavioral: Intensive Info-Motivation-Behavioral Skills Intervention
- 5 (Experimental): Brief Informational Intervention + Intensive Informational Intervention
  Interventions: Behavioral: Brief Informational Intervention; Behavioral: Intensive Informational Intervention
- 6 (Experimental): Brief Informational Intervention + Intensive Information-Motivation-Behavioral Skills Intervention
  Interventions: Behavioral: Brief Informational Intervention; Behavioral: Intensive Info-Motivation-Behavioral Skills Intervention

INTERVENTIONS:
Behavioral: Brief Motivational Intervention — 15-20 minute, motivational one-on-one counseling
  Arms: 1; 3; 4
Behavioral: Brief Informational Intervention — 15 minute informational DVD on safer sex
  Arms: 2; 5; 6
Behavioral: Intensive Informational Intervention — 4-hour, information-only intensive group workshop
  Arms: 3; 5
Behavioral: Intensive Info-Motivation-Behavioral Skills Intervention — 4-hour, intensive group workshop with emphasis on motivation and skills
  Arms: 4; 6

SUMMARY:
This study will determine the effectiveness of a two-step HIV prevention program in reducing risky sexual practices and decreasing the incidence of sexually transmitted diseases (STDs).

DETAILED DESCRIPTION:
Numerous factors influence one's sexual choices, including social support and pressure, internal feelings and beliefs, and knowledge about the subject. Data indicate that people who are well-informed about the risks associated with certain sexual behaviors are more likely to protect themselves than those who are less informed. This study will determine whether an intervention comprising information, motivation, and behavioral skills components is more effective than an information-only workshop in changing sexual behavior for HIV prevention.

At study entry, participants will undergo a physical exam, various STD tests, and a rapid HIV test, which can provide test results within several hours. While waiting for their test results at the study clinic, participants will complete a computerized questionnaire assessing their thoughts, feelings, and behaviors regarding sexual activities. Participants will also be exposed to one of two brief health promotion interventions: a motivational, one-on-one counseling session or a DVD on safer sex. After receiving their test results, participants will be asked to complete a brief postassessment questionnaire about their attitudes toward their test results and the intervention.

Two-thirds of the participants will then be invited to attend an intensive, 4-hour safer sex workshop. These participants will be randomly assigned to one of two workshops: an information-only workshop or a workshop that includes information, motivation, and behavioral skills components. Participants who choose not to participate in the workshop will complete the study after receiving their STD and HIV test results. Participants who participate in the workshop will return to the clinic at 3, 6, and 12 months after the workshop to complete another questionnaire about sexual behaviors and give a urine sample for STD testing.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis or symptoms of an STD within 3 months prior to study entry OR have had unprotected vaginal or anal intercourse with one or more of the following: two or more sexual partners, a partner with two or more partners, an anonymous partner, an injection drug-using partner, or a partner with an STD
* Able to understand English

Exclusion Criteria:

* Psychosis or impaired mental status that would prevent participant from providing informed consent
* Have been tested for HIV within 3 months prior to study entry
* HIV infected

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1554 (Actual)
Dates: Start 2004-03; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Sexual behavior | 12 months

SECONDARY OUTCOMES:
STD incidence | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael P. Carey, PhD, Principal Investigator — Syracuse University
Locations (1):
- Syracuse University, Syracuse, New York, United States